CLINICAL TRIAL: NCT01695655
Title: Neovascularization Patterns in Corneal Graft Rejection
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roni Shtein, Assistant Professor, University of Michigan
Other Study IDs: Neovasc-6281
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Corneal Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PKP: Subjects undergoing penetrating keratoplasty

SUMMARY:
Corneal transplantation is the most commonly performed human tissue transplant worldwide. Over 40,000 corneal transplants occur in the US each year. .

This study will determine specific corneal neovascularization (CN) patterns in human corneal allograft recipients to determine the characteristics that worsen the prognosis for graft survival. We will test the hypothesis that specific characteristics of CN are prognostic for corneal allograft rejection.

DETAILED DESCRIPTION:
The investigators hope to enroll 240 subjects into the study. These patients will be enrolled prior to penetrating keratoplasty. They will be examined by the full protocol preoperatively, and postoperatively at 1 week, 1, 3, 6, 12, 18, and 24 months. During these visits slit lamp biomicroscopy will be used to study CN patterns, and take slit lamp photographs if there is any neovascularization detected, permitting us to develop algorithms of CN characteristics that are predictive for corneal allograft rejection and failure. The corneal tissue removed during these patients' surgeries will be evaluated histopathologically to identify inflammation and neovascularization to confirm and compare to what is seen clinically. There will be two short questionnaires conducted at each visit to assess stress levels.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for corneal transplant

Exclusion Criteria:

* previous corneal transplant

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: subjects with indications of corneal transplant
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2007-11; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Corneal graft rejection | 0 to 2 years after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Roni Shtein, MD, MS, Principal Investigator — University Of Michigam Kellogg Eye Center
Locations (1):
- Kellogg Eye Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No